CLINICAL TRIAL: NCT01020994
Title: Explorative, Double-blind, Randomized, Controlled Multi-center Phase II Study to Evaluate the Efficacy and Safety of Topically Applied LAS41003 Once Daily Versus LAS189962 and LAS189961 in the Treatment of Superficial Infected Eczema
Brief Title: Efficacy and Safety of LAS41003 in the Treatment of Superficial Infected Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Head of Global Clinical Development, Almirall Hermal GmbH
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H 552 000 - 0911; EudraCT: 2009-011931-11
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Eczema
Keywords: Superficial infected eczema; Superinfected eczema
MeSH Terms: conditions — Eczema | interventions — octenidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- LAS41003 (Experimental)
  Interventions: Drug: LAS41003
- LAS189962 (Active Comparator)
  Interventions: Drug: LAS189962
- LAS189961 (Active Comparator)
  Interventions: Drug: LAS189961

INTERVENTIONS:
Drug: LAS41003 — Once daily, topically
  Arms: LAS41003
Drug: LAS189962 — Once daily, topically
  Arms: LAS189962
Drug: LAS189961 — Once daily, topically
  Arms: LAS189961

SUMMARY:
The aim of the study is to determine the efficacy and safety of topical application of LAS41003 in comparison to LAS189962 and LAS189961 in the treatment of superinfected eczema.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed super-infected or impetiginized eczema

Exclusion Criteria:

* Patients who have general signs of systemic infections like fever, malaise, lymphangitis or swollen lymph nodes and / or need systemic antibiotic treatment
* Patients who have a bacterial skin infection which, due to depth and severity, could not be appropriately treated with a topical antimicrobial or antiseptic medication
* Diagnose of the following disease:

  * Known active tuberculosis or any history of past tuberculosis of skin
  * Suspected or proven parasitic infection of the treatment site (e.g. scabies)
  * Psoriasis
  * Suspected or proven viral infection of skin (e.g. Herpes)
* Localization of the superficial infected eczema:

  * Palms of the hands
  * Sole of a foot
  * Face
* Have received any topical treatment with antibiotics, antimycotics, immunomodulators and corticosteroid preparations within the last 2 weeks before treatment with IMP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Combination of clinical and microbial treatment success | Day 14

SECONDARY OUTCOMES:
Safety:Physical examination at EoT, AEs/SAEs during the entire study | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, MBA, Study Director — Almirall Hermal GmbH
Locations (1):
- Investigational Site, Bochum, Germany